CLINICAL TRIAL: NCT04605692
Title: Attitudes and Predictive Factors of Psychological Distress and Occupational Burnout Among Dentists During COVID-19 Pandemic in Turkey
Brief Title: Evaluation of Occupational Burnout and Stress Among Dentists in Covid-19 Pandemic
Acronym: MBI
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Merve Özarslan, Research Assissant Dr., Akdeniz University
Other Study IDs: KAEK- 590
Record Dates: First submitted 2020-10-26; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Burnout; COVID-19; Dentistry; Filiation; Pandemic
MeSH Terms: conditions — Burnout, Psychological; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to evaluate the factors affecting the ability and willingness of dentists to work during the COVID-19 pandemic and the effect of this situation on occupational burnout. A 51-question survey, including demographic and pandemic questions and the Maslach Burnout Inventory (MBI), was used as a data collection method and administered to dentists in Turkey via the internet in two stages. A link to the survey (onlineanketler.com) was sent to the participants by e-mail or social media (WhatsApp©). A total of 706 participants were included in the study. The second stage of the survey only applied to dentists who are assigned within the scope of COVID-19 measures in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* All dentist working during the COVID-19 outbreak
* Accepted electronically to participate in our study
* Completed and submitted our electronic questionnaires successfully

Exclusion Criteria:

* Non-dentists
* Did not accept electronically to participate in our study
* Did not complete not submitted our electronic questionnaires successfully

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants included dentists dealing with COVID-19 patients vs. those who are not dealing with COVID-19 patients from hospitals and health centers inside Turkey, totaly 706.
  Our questionnaires were used to assess their mental health by measuring burnout and stress levels. Participants' socio-demographic data such as age, gender, profession, marital state, years of experience, weekly working hours were collected.
Sampling Method: Probability Sample
Enrollment: 706 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
706 of participants' burnout (MBI) and stress levels during the Covid 19 pandemic process assessed with survey. | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz Üniversitesi, Antalya, Konyaaltı, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozarslan M, Caliskan S. Attitudes and predictive factors of psychological distress and occupational burnout among dentists during COVID-19 pandemic in Turkey. Curr Psychol. 2021;40(7):3113-3124. doi: 10.1007/s12144-021-01764-x. Epub 2021 Apr 29. PMID 33948050